CLINICAL TRIAL: NCT07343453
Title: A Single-Arm, Phase II Study to Evaluate the Efficacy and Safety of Sacituzumab Tirumotecan in Second-Line and Subsequent Treatments for Advanced Thymic Epithelial Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Hou, Professor of Medicine, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-864-02
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Thymic Epithelial Tumors; Advanced Stage; Second-line Therapy

STUDY DESIGN:
Intervention Model Description: Sacituzumab Tirumotecan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Tirumotecan (Experimental): Sacituzumab Tirumotecan, 5 mg/kg, iv. drip, D1 and D15, Q4W. Treatment will continue until disease progression (as defined by loss of clinical benefit), intolerable toxicity, patient withdrawal, or meeting other protocol-specified discontinuation criteria.
  Interventions: Drug: Sacituzumab tirumotecan

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — Sacituzumab Tirumotecan is an antibody-drug conjugate (ADC) composed of a humanized anti-TROP2 monoclonal antibody of the IgG1 class covalently linked to the cytotoxic payload KL610023, a topoisomerase I inhibitor. Its mechanism of action involves: (1) specific binding of the antibody to Trop-2 on the tumor cell membrane, followed by internalization; (2) lysosomal degradation leading to the release of SN-38, which induces DNA double-strand breaks; and (3) a bystander effect that kills adjacent Trop-2-negative cells.

SUMMARY:
This is a single-arm, phase II study to evaluate the efficacy and safety of Sacituzumab Tirumotecan, a TROP2-directed antibody-drug conjugate, in patients with advanced thymic epithelial tumors who have received second-line or later therapy.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of Sacituzumab Tirumotecan, a TROP2-directed antibody-drug conjugate, in patients with advanced thymic epithelial tumors who have received second-line or later therapy. The study is designed as a prospective, single-arm, phase II clinical trial. Eligible patients must meet the inclusion/exclusion criteria, have received prior systemic therapy, and have a pathological diagnosis of advanced thymic epithelial tumor. Enrolled patients will receive Sacituzumab Tirumotecan at a dose of 5 mg/kg via intravenous infusion. Treatment cycles repeat every 4 weeks, with administration on Day 1 and Day 15 of each cycle. Treatment will continue until disease progression (as defined by loss of clinical benefit), intolerable toxicity, patient withdrawal, or meeting other protocol-specified discontinuation criteria. The primary endpoint of this study is the Objective Response Rate (ORR), defined as the proportion of patients achieving a confirmed Complete Response (CR) or Partial Response (PR) as their best overall response, assessed according to RECIST version 1.1. Secondary endpoints include Progression-Free Survival (PFS), Disease Control Rate (DCR), Duration of Response (DOR), Overall Survival (OS), incidence of Adverse Events (AEs), and Quality of Life (QoL) assessments. Following treatment discontinuation, subjects will enter a follow-up phase consisting of safety follow-up and survival follow-up, with survival status assessed every 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced (unresectable or metastatic) thymic epithelial tumor confirmed by histology or cytology.
2. Progress after receiving at least first-line systemic therapy (chemotherapy or immune checkpoint inhibitor).
3. According to RECISTv1.1 standard, there is at least one measurable lesion.
4. No central nervous system metastasis or stable brain metastasis after treatment (asymptomatic and hormone withdrawal for ≥4 weeks).
5. Age > 18 years old, male or female.
6. ECOG (Performance status, PS) score 0-1.
7. Expected survival time ≥12 weeks.
8. Organ function compliance (confirmed by laboratory examination within 14 days before treatment): Bone marrow function: I. Neutrophils ≥ 1500× 109/L; Ii. Platelets ≥ 100× 109/L; Iii. hemoglobin > 90g/l; Renal function: I. Serum creatinine ≤1.5×ULN or creatinine clearance rate (CrCl). ≥50mL/min； Ii. Urine protein < 2+or 24H urine protein quantitative < <1.0g；; Liver function: I, AST or ALT ≤ 3× ULN; For patients with liver metastasis, it can ≤5*ULN； Ii. Total bilirubin ≤1.5×ULN, and liver metastasis patients ≤ 3× ULN; Iii: serum albumin (ALB) ≥ 28g/l; Coagulation function: NR or APTT≤1.5×ULN；; Cardiac function: Left ejection fraction (LEFF) ≥ 50%.
9. Before making any evaluation related to the study, the subjects must understand and volunteer. Sign the informed consent form and voluntarily comply with other requirements of the study.
10. Female subjects with reproductive function must be treated within 3 days before the first medication. Urine or serum pregnancy test (if the result of urine pregnancy test cannot be confirmed as negative, serum pregnancy test is needed, and the serum pregnancy result shall prevail). If a fertile woman has sex with an unsterilized male partner, the subjects agree to continue using contraception and avoid breastfeeding during the medication.
11. Male subjects are willing to agree to continue using contraception during the medication.

Exclusion Criteria:

1. Previously received targeted drug therapy with Lucasatuzumab.
2. Have received any drug therapy targeting topoisomerase I in the past, including antibody-coupled drug (ADC) therapy.
3. Patients with grade 3-4 interstitial lung disease.
4. Subjects known to have meningeal metastasis, brain stem metastasis, spinal cord metastasis and/or compression, active or brain metastasis without local treatment. 5.Subjects with brain metastases who have previously received local treatment can participate in the study if they are clinically stable for at least 4 weeks before the first administration of the study treatment and do not need to use corticosteroids or anticonvulsants for at least 14 days before the first administration; For the subjects with brain metastases first discovered during screening, if they receive local treatment (such as radiotherapy), they must have imaging evidence to show that the brain metastases have not progressed for at least 4 weeks from the first imaging diagnosis of brain metastases, and they can only enter the group after confirming that the brain metastases are stable.
5. Patients with previous malignant tumors (except skin malignant tumors other than melanoma, and carcinoma in situ in the following parts [bladder, stomach, colorectal cancer, endometrium, cervix, melanoma or breast]) cannot be included in this study. However, if the malignant tumor has achieved complete remission for five years or more, and no additional anti-tumor treatment is needed during this study, it can be included in the study.
6. Myocardial infarction and uncontrolled arrhythmia occurred within 6 months before the first administration (including QTc interval ≥450ms for men and ≥ 470 ms for women) (QTc interval is calculated by Fridericia formula); Or grade III-IV cardiac insufficiency according to NYHA standard or left ventricular ejection fraction < 50% by color Doppler echocardiography.
7. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage. Only a small amount of pleural effusion, a small amount of ascites and a small amount of pericardial effusion without clinical symptoms shown by imaging can be included in the group.
8. Subjects with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcer, gastrointestinal perforation, abdominal abscess or acute gastrointestinal bleeding.
9. Patients with active hepatitis B, hepatitis C, tuberculosis and syphilis or other serious infections with poor clinical control.
10. HIV positive or diagnosed with acquired immunodeficiency disease (AIDS).
11. Known allergic to the study drug or any of its components (including polysorbate -20), known history of severe hypersensitivity to other monoclonal antibodies (NCI-CTCAE5.0 grade is greater than grade 3).
12. Before the first administration, he was receiving long-term systemic corticosteroid therapy of > 10mg of prednisone or equivalent dose of systemic corticosteroid therapy or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy. Subjects who need bronchodilators, inhaled or topical steroids or local steroid injections, and who are used as preventive drugs for hypersensitivity (such as drugs before CT examination) may be admitted into the group.
13. Known history of hereditary bleeding tendency disease or coagulation dysfunction.
14. Pregnant or lactating women.
15. During the screening before the first administration, the condition deteriorated rapidly, such as serious changes in physical state.
16. The researcher thinks that the patient can't finish the study medically, psychologically or physically or can't understand the information in the patient manual.
17. Those who have been vaccinated with live or attenuated vaccines within 28 days before the first administration or have plans to vaccinate such vaccines during the study period; However, inactivated virus vaccines for seasonal influenza are allowed to be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-12-22 (Estimated); Study Completion 2029-12-22 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | Within one year after starting treatment.
  ORR, per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression free survival （PFS） | Within two year after the first treatment
  The time interval from the first dose of study medication to the first record of disease progression or death from any cause, whichever occurred first.
Disease control rate (DCR) | Within one year after starting treatment.
  The proportion of subjects who achieved the best total efficacy was to confirm CR or PR or SD (according to iRECIST).
Duration of remission (DOR) | Within one year after starting treatment.
  The time from the first record of confirmed remission (CR or PR) to the first record of disease progression (according to irecist) or death due to any cause, whichever occurs first.
Overall survival (OS) | Assessed from enrollment to death or last known survival, up to 4 years post-enrollment.
  OS is defined as the time from the first administration of the study drug until the date of death from any cause. For subjects who are alive at the data cutoff, censoring will occur at the last known date of survival. Subjects with no follow-up information provided will be censored on the date of enrollment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tagawa ST, Balar AV, Petrylak DP, Kalebasty AR, Loriot Y, Flechon A, Jain RK, Agarwal N, Bupathi M, Barthelemy P, Beuzeboc P, Palmbos P, Kyriakopoulos CE, Pouessel D, Sternberg CN, Hong Q, Goswami T, Itri LM, Grivas P. TROPHY-U-01: A Phase II Open-Label Study of Sacituzumab Govitecan in Patients With Metastatic Urothelial Carcinoma Progressing After Platinum-Based Chemotherapy and Checkpoint Inhibitors. J Clin Oncol. 2021 Aug 1;39(22):2474-2485. doi: 10.1200/JCO.20.03489. Epub 2021 Apr 30. PMID 33929895
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Gomez Pardo P, Jhaveri KL, Delaney R, Valdez T, Wang H, Motwani M, Yoon OK, Verret W, Tolaney SM. Overall survival with sacituzumab govitecan in hormone receptor-positive and human epidermal growth factor receptor 2-negative metastatic breast cancer (TROPiCS-02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1423-1433. doi: 10.1016/S0140-6736(23)01245-X. Epub 2023 Aug 23. PMID 37633306
- [Background] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206
- [Background] Lombardi P, Filetti M, Falcone R, Altamura V, Paroni Sterbini F, Bria E, Fabi A, Giannarelli D, Scambia G, Daniele G. Overview of Trop-2 in Cancer: From Pre-Clinical Studies to Future Directions in Clinical Settings. Cancers (Basel). 2023 Mar 13;15(6):1744. doi: 10.3390/cancers15061744. PMID 36980630
- [Background] Dum D, Taherpour N, Menz A, Hoflmayer D, Volkel C, Hinsch A, Gorbokon N, Lennartz M, Hube-Magg C, Fraune C, Bernreuther C, Lebok P, Clauditz TS, Jacobsen F, Sauter G, Uhlig R, Wilczak W, Steurer S, Minner S, Marx AH, Simon R, Burandt E, Krech T, Luebke AM. Trophoblast Cell Surface Antigen 2 Expression in Human Tumors: A Tissue Microarray Study on 18,563 Tumors. Pathobiology. 2022;89(4):245-258. doi: 10.1159/000522206. Epub 2022 Apr 27. PMID 35477165
- [Background] Ardeshir-Larijani F, Maniar R, Goyal S, Loehrer PJ, Hou T, DeBrock V, Mesa H. Trop-2 Expression and Its Impact on Survival in Thymic Epithelial Tumors: Brief Report. Clin Lung Cancer. 2024 Mar;25(2):180-185.e1. doi: 10.1016/j.cllc.2024.01.001. Epub 2024 Jan 2. No abstract available. PMID 38242729
- [Background] Kurokawa K, Asao T, Hayashi T, Kishikawa S, Kanamori K, Shukuya T, Miyashita Y, Nakamura I, Miyawaki T, Kanemaru R, Mimori T, Mitsuishi Y, Tajima K, Shimada N, Takahashi F, Takamochi K, Suzuki K, Takahashi K. Trophoblast Cell Surface Antigen 2 Expression in Thymic Carcinoma: Brief Report. JTO Clin Res Rep. 2024 May 29;5(7):100693. doi: 10.1016/j.jtocrr.2024.100693. eCollection 2024 Jul. PMID 39034967
- [Background] Yeung V, Zaemes J, Yeh J, Giancarlo C, Ahn J, Reuss JE, Kallakury BV, Liu SV, Duttargi A, Khan G, Kim C. High levels of expression of Trop-2 in thymic epithelial tumors. Lung Cancer. 2023 Oct;184:107324. doi: 10.1016/j.lungcan.2023.107324. Epub 2023 Aug 9. PMID 37573703
- [Background] Huang Q, Zhu L, Liu Y, Zhang Y. Thymic epithelial tumor medical treatment: A narrative review. Biochim Biophys Acta Rev Cancer. 2024 Sep;1879(5):189167. doi: 10.1016/j.bbcan.2024.189167. Epub 2024 Aug 6. PMID 39117091
- [Background] Girard N, Ruffini E, Marx A, Faivre-Finn C, Peters S; ESMO Guidelines Committee. Thymic epithelial tumours: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v40-55. doi: 10.1093/annonc/mdv277. No abstract available. PMID 26314779
- [Background] Li Y, Jiang A, Zhao Y, Shi C, Ma Y, Fu X, Liang X, Tian T, Ruan Z, Yao Y. A novel risk classifier for predicting the overall survival of patients with thymic epithelial tumors based on the eighth edition of the TNM staging system: A population-based study. Front Endocrinol (Lausanne). 2022 Dec 6;13:1050364. doi: 10.3389/fendo.2022.1050364. eCollection 2022. PMID 36561557
- [Background] Marx A, Willcox N, Leite MI, Chuang WY, Schalke B, Nix W, Strobel P. Thymoma and paraneoplastic myasthenia gravis. Autoimmunity. 2010 Aug;43(5-6):413-27. doi: 10.3109/08916930903555935. PMID 20380583
- [Background] Cheng M, Anderson MS. Thymic tolerance as a key brake on autoimmunity. Nat Immunol. 2018 Jul;19(7):659-664. doi: 10.1038/s41590-018-0128-9. Epub 2018 Jun 20. PMID 29925986
- [Background] Kurokawa K, Shukuya T, Greenstein RA, Kaplan BG, Wakelee H, Ross JS, Miura K, Furuta K, Kato S, Suh J, Sivakumar S, Sokol ES, Carbone DP, Takahashi K. Genomic characterization of thymic epithelial tumors in a real-world dataset. ESMO Open. 2023 Oct;8(5):101627. doi: 10.1016/j.esmoop.2023.101627. Epub 2023 Sep 12. PMID 37703595
- [Background] Radovich M, Pickering CR, Felau I, Ha G, Zhang H, Jo H, Hoadley KA, Anur P, Zhang J, McLellan M, Bowlby R, Matthew T, Danilova L, Hegde AM, Kim J, Leiserson MDM, Sethi G, Lu C, Ryan M, Su X, Cherniack AD, Robertson G, Akbani R, Spellman P, Weinstein JN, Hayes DN, Raphael B, Lichtenberg T, Leraas K, Zenklusen JC; Cancer Genome Atlas Network; Fujimoto J, Scapulatempo-Neto C, Moreira AL, Hwang D, Huang J, Marino M, Korst R, Giaccone G, Gokmen-Polar Y, Badve S, Rajan A, Strobel P, Girard N, Tsao MS, Marx A, Tsao AS, Loehrer PJ. The Integrated Genomic Landscape of Thymic Epithelial Tumors. Cancer Cell. 2018 Feb 12;33(2):244-258.e10. doi: 10.1016/j.ccell.2018.01.003. PMID 29438696
- [Background] Marx A, Chan JKC, Chalabreysse L, Dacic S, Detterbeck F, French CA, Hornick JL, Inagaki H, Jain D, Lazar AJ, Marino M, Marom EM, Moreira AL, Nicholson AG, Noguchi M, Nonaka D, Papotti MG, Porubsky S, Sholl LM, Tateyama H, Thomas de Montpreville V, Travis WD, Rajan A, Roden AC, Strobel P. The 2021 WHO Classification of Tumors of the Thymus and Mediastinum: What Is New in Thymic Epithelial, Germ Cell, and Mesenchymal Tumors? J Thorac Oncol. 2022 Feb;17(2):200-213. doi: 10.1016/j.jtho.2021.10.010. Epub 2021 Oct 22. PMID 34695605
- [Background] Xu C, Zhang Y, Wang W, Wang Q, Li Z, Song Z, Wang J, Yu J, Liu J, Zhang S, Cai X, Wu M, Zhan P, Liu H, Lv T, Miao L, Min L, Li J, Liu B, Yuan J, Jiang Z, Lin G, Chen X, Pu X, Rao C, Lv D, Yu Z, Li X, Tang C, Zhou C, Zhang J, Guo H, Chu Q, Meng R, Liu X, Wu J, Hu X, Fang M, Zhou J, Zhu Z, Chen X, Pan W, Pang F, Zhou Y, Jian Q, Wang K, Wang L, Zhu Y, Yang G, Lin X, Cai J, Liang L, Feng H, Wang L, Du Y, Yao W, Shi X, Niu X, Yuan D, Yao Y, Huang J, Zhang Y, Sun P, Wang H, Ye M, Wang D, Wang Z, Hao Y, Wang Z, Wan B, Lv D, Yu G, Li A, Kang J, Zhang J, Zhang C, Chen H, Shi L, Ye L, Wang G, Wang Y, Gao F, Zhou W, Hu C, Wei J, Li B, Li Z, Li Y, Liu Z, Yang N, Wu L, Wang Q, Huang W, Hong Z, Wang G, Fang M, Fang Y, Zhu X, Du K, Ji J, Shen Y, Zhang Y, Ma S, Song Y, Lu Y, Liu A, Fang W, Zhong W. Chinese expert consensus on the diagnosis and treatment of thymic epithelial tumors. Thorac Cancer. 2023 Apr;14(12):1102-1117. doi: 10.1111/1759-7714.14847. Epub 2023 Mar 16. PMID 36924056
- [Background] Gerber TS, Strobl S, Marx A, Roth W, Porubsky S. Epidemiology of thymomas and thymic carcinomas in the United States and Germany, 1999-2019. Front Oncol. 2024 Jan 9;13:1308989. doi: 10.3389/fonc.2023.1308989. eCollection 2023. PMID 38264756